CLINICAL TRIAL: NCT00904475
Title: A Prospective, Prospective, Double-blind, Randomized, Placebo-Controlled, Pilot Study of the Efficacy and Safety of Lidoderm Patch in the Treatment of Low Back Pain
Brief Title: Pilot Study of the Efficacy and Safety of Lidoderm Patch in the Treatment of Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, Clinical R&D, Endo Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3220-011
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Lidoderm

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1- Lidoderm® (Experimental): Lidoderm (lidocaine patch 5%), up to three patches applied topically once daily (q24h) to the area of maximal peripheral pain
  Interventions: Drug: Lidoderm®
- 2-Placebo (Placebo Comparator): Matching placebo, up to three patches applied topically once daily (q24h) to the area of maximal peripheral pain
  Interventions: Drug: Lidoderm®

INTERVENTIONS:
Drug: Lidoderm® — Eligible patients were randomized equally to one of two groups: lidocaine patch 5% or matching placebo patch. During the 6-week treatment period, patients used up to three patches daily applied q24h.
  Other Names: Lidocaine patch 5%
  Arms: 1- Lidoderm®
Drug: Lidoderm® — Eligible patients were randomized equally to one of two groups: lidocaine patch 5% or matching placebo patch. During the 6-week treatment period, patients used up to three patches daily applied q24h.
  Other Names: Lidocaine patch 5%
  Arms: 2-Placebo

SUMMARY:
Patients with moderate to severe chronic Low Back Pain (LBP) despite current analgesic treatment participated in a Phase IV clinical trial to evaluate the analgesic efficacy of the lidocaine patch 5% compared to placebo in treating moderate to severe chronic LBP.

ELIGIBILITY:
Inclusion Criteria:

1. Were currently experiencing moderate/severe pain despite current analgesic treatment
2. Had daily moderate-to-severe LBP for at least 3 months duration
3. Had a mean daily pain intensity score of >6 on a 0 to 10 scale, with 0 being no pain and 10 being pain as bad as the patients have ever imagined (Question 5 of BPI) during the baseline week; patients had to complete daily diary assessments at least 5 of 7 days during the baseline week

Exclusion Criteria:

1. Had a history of greater than one back surgery, or one back surgery within 3 months of study entry
2. Had severe spinal stenosis
3. Had chronic back pain of >12 months duration with an undefined spinal diagnosis
4. Had radicular symptoms with radiation into the thigh or below (i.e., knee, calf, foot, etc.)
5. Had received an epidural steroid/local anesthetic injection within 2 weeks prior to study entry
6. Had received trigger point injections within 2 weeks prior to study entry
7. Had received Botulinum Toxin Injections for LBP within 3 months prior to study entry
8. Were taking a lidocaine-containing product that could not be discontinued while receiving study medication
9. Were taking class 1 anti-arrhythmic drugs (e.g., mexiletine, tocainide)
10. Had received Lidoderm for LBP in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-04; Primary Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Mean change in average daily pain intensity (BPI Question 5) from baseline week to the final week of treatment (primary endpoint) | Visit - V2 (Day 0), V3 (Day 7), V4 (Day 14), V5 (Day 28), V6/EOS (Day 42)

SECONDARY OUTCOMES:
Mean change from baseline to Week 2 and Week6/EOS in average daily pain intensity (BPI Question 5)
Pain relief (BPI Question 8)
Mean change from baseline to Week 2 and Week 6 in Pain Quality Assessment Scale (PQAS)
Patient and Investigator Global Impression of Pain Relief at Week 6
QoL: Change from baseline to Week 6 in pain interference with QoL (BPI Question 9) and Profile of Mood States (POMS)
Safety assessments included AEs, discontinuations as a result of AEs, clinical laboratory tests, vital signs, physical examination, plasma lidocaine levels, dermal assessments and sking sensory testing

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Study Director — Endo Pharmaceuticals
Locations (6):
- United States (6):
  - Birmingham, Alabama
  - Hueytown, Alabama
  - Phoenix, Arizona
  - Mill Valley, California
  - Allentown, Pennsylvania
  - Salt Lake City, Utah